CLINICAL TRIAL: NCT05692219
Title: Comparative Efficacy of Self-Help Multicomponent Lifestyle Medicine Intervention and Cognitive Behavioral Therapy for Depressive Symptoms: A Pilot Randomized Controlled Trial
Brief Title: Comparative Efficacy of Self-Help Multicomponent Lifestyle Medicine Intervention and Cognitive Behavioral Therapy for Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSY027
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Depression
Keywords: Lifestyle Medicine; Cognitive Behavioural Therapy; Self-help
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle medicine (Experimental): The booklet-delivered multicomponent lifestyle medicine intervention includes six weekly sessions (i.e., participants are anticipated to access the intervention every day for 42 days) that are related to the following topics: (a) lifestyle psychoeducation, (b) exercise, (c) nutritional recommendations, (d) stress management, (e) sleep management, and (f) motivation and goal-setting techniques.
  Interventions: Behavioral: Lifestyle medicine
- Cognitive behavioural therapy (Active Comparator): The booklet-delivered self-help CBT includes six weekly sessions (i.e., participants are anticipated to access the intervention every day for 42 days) that are related to psychoeducation of depression, cognitive behavioural techniques( e.g. behavioral activation, cognitive restructuring), stress management, mindfulness, goal-setting, and/or positive psychology.
  Interventions: Behavioral: Cognitive behavioral therapy
- Waitlist control (No Intervention): Participants in the waitlist control group will be asked to maintain their typical activities during the trial period, and they will be given the lifestyle medicine booklet or CBT booklet based on their preference following the completion of the 3-month follow-up assessment (Week 19).

INTERVENTIONS:
Behavioral: Lifestyle medicine — 6 weeks booklet-delivered multicomponent lifestyle medicine intervention
  Arms: Lifestyle medicine
Behavioral: Cognitive behavioral therapy — 6 weeks booklet-delivered self-help cognitive behavioral therapy
  Arms: Cognitive behavioural therapy

SUMMARY:
The objective of this proposed pilot randomized controlled trial is to examine the efficacy of self-help multicomponent lifestyle medicine intervention and cognitive behavioral therapy relative to a wait-list control group for alleviating depressive symptoms among Hong Kong Chinese adults.

DETAILED DESCRIPTION:
This study will serve as a pioneering attempt to investigate the comparative efficacy of self-help multicomponent lifestyle medicine intervention and cognitive behavioral therapy for reducing depressive symptoms. The proposed study will pave the way for future intervention development and provide the evidence base for the integration of lifestyle-based interventions into the current treatment model.

Prior to all study procedures, eligible participants will be required to complete an online informed consent via an in-house smartphone application, Longitudinax Pro. Around 90 eligible participants aged 18 or above with a Patient Health Questionnaire-9 total score of 10 or higher will be randomly assigned to either self-help multicomponent lifestyle medicine intervention (LM), self-help CBT (CBT), or the waitlist control group (WL) in a ratio of 1:1:1 by an independent statistician. Participants in the LM and CBT groups will receive a booklet-delivered multicomponent lifestyle medicine intervention and CBT for depressive symptoms, respectively. Both interventions comprise 6 weekly 60-minute sessions and daily homework activities according to instructions in the booklet (details can be found in "Arms and Interventions"). For both LM and CBT groups, a follow-up phone call (approximately 15 minutes) will be made every two weeks to encourage participants to adhere to the intervention. Participants in the WL group will be asked to maintain their typical activities during the trial period, and they will be given access to either the booklet-delivered multicomponent lifestyle medicine intervention or booklet-delivered CBT following the 3-month post-intervention follow-up. The primary outcome of interest will be depressive symptoms. The secondary outcomes will include anxiety symptoms, perceived insomnia severity, health-promoting behaviors, quality of life, functional impairment, and intervention evaluation at immediate post-intervention and 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged 18 or above
* Able to read Chinese and write in Chinese or English
* Have a Patient Health Questionnaire-9 (PHQ-9) total score of 10 or higher indicating at least moderate level of depressive symptoms
* Willing to provide informed consent and comply with the trial protocol
* Have an Internet-enabled mobile device (iOS or Android operating system) (for data collection purposes)

Exclusion Criteria:

* Received psychotherapy for depression and/or insomnia in the past 6 months
* A change in psychotropic drugs or over-the-counter medications that target depression and/or insomnia within 2 weeks before the baseline assessment
* A PHQ-9 item-9 score equal to or higher than 2, indicating a moderate level of suicidal risk that requires active crisis management (referral information to professional mental health services will be provided)
* Currently participating in another interventional study that may potentially improve mental health
* Pregnancy
* Self-disclosure of having unsafe conditions for which physical activity or a change in diet was contraindicated by physicians or other health professionals (e.g., dietitian)
* Self-disclosure of a diagnosis of any major psychiatric, medical, or neurocognitive disorders that make participation unsuitable or interfere with the adherence to the interventions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in The Patient Health Questionnaire (PHQ-9) | Baseline, immediate post-intervention, and 3-month post-intervention
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in The Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediate post-intervention, and 3-month post-intervention
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-intervention, and 3-month post-intervention
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediate post-intervention, and 3-month post-intervention
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in The Short Multidimensional Inventory Lifestyle Evaluation (SMILE) | Baseline, immediate post-intervention, and 3-month post-intervention
  The SMILE is a 43-item self-report questionnaire designed to measure 7 aspects of lifestyle, which included diet and nutrition (7-item), substance use (4-item), exercise (3-item), stress management (10-item), sleep management (5- item), social support (10-item), and environmental exposures (4-item). Each item is rated on a 4-point Likert scale. The possible response categories of each item are always (4), several days (3), seldom (2), and never (1). For items 3-4, 8-11, 21, 29, and 40-41, they will be reverse scored. The total score of a lifestyle aspect equals the sum of the respected item score, while the overall lifestyle pattern score can be calculated by summing up the 43-item scores. The higher the score, the better the lifestyle pattern.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediate post-intervention, and 3-month post-intervention
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediate post-intervention, and 3-month post-intervention
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from a short form of the International Physical Activity Questionnaire - Chinese version a short form of the IPAQ-C.
Change in the Treatment Acceptability and Adherence Scale (TAAS) | Baseline and immediate post-intervention
  TAAS is a self-reported, ten-item questionnaire that is rated by a seven-point Likert scale from 1 to 7, and it aims at evaluating the clients' attitude toward the treatment sessions by four domains, including acceptability, adherence, drop-out, and distress. Specific wording referencing "anxiety" was changed to refer to "depression".
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-intervention
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success. Specific wording referencing "anxiety" was changed to refer to "depression".
Self-developed survey | Baseline
  The self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence), substance use, body mass index (BMI), rest-activity pattern, and social rhythms, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Yan-Yee Ho, PhD, Study Chair — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No